CLINICAL TRIAL: NCT01313702
Title: Effect of Polipill on Patients at High Cardiovascular Risk : a Randomized Controlled Trial
Brief Title: Single Pill to Avert Cardiovascular Events
Acronym: SPACE
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital do Coracao (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IEP001/2011
Record Dates: First submitted 2011-03-10; First posted 2011-03-14 (Estimated); Last update posted 2022-09-21 (Actual); Status verified 2012-03

CONDITIONS: Cardiovascular Disease
Keywords: polypill, compliance, cardiovascular disease
MeSH Terms: conditions — Cardiovascular Diseases; Patient Compliance | interventions — Lisinopril; Simvastatin; Atenolol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- polipillV1 (Experimental): poli pill version 1: aspirin 75mg, simvastatin 40mg, lisinopril 10mg, atenolol 50mg
  Interventions: Drug: polipillV1
- polipillV2 (Experimental): Polipill versão2: aspirin 75mg, simvastatin 40mg, lisinopril 10mg, hydrochlorothiazide 12.5mg.
  Interventions: Drug: polipillV2
- usual care (Active Comparator)
  Interventions: Drug: usual care

INTERVENTIONS:
Drug: polipillV1 — polipill version 1: aspirin 75mg, simvastatin 40mg, lisinopril 10mg, atenolol 50mg
  Other Names: no other name
  Arms: polipillV1
Drug: polipillV2 — Polipill version 2: aspirin 75mg, simvastatin 40mg, lisinopril 10mg, hydrochlorothiazide 12.5mg.
  Other Names: no other name
  Arms: polipillV2
Drug: usual care — the drugs used in clinical practice, defined by physician
  Other Names: lisinopril; simvastatin; atenolol; hidrochlorotiazide; acetylsalicilic acid
  Arms: usual care

SUMMARY:
The purpose of this study is to determine whether a polipill improved the compliance with treatment compared to usual care that use two or more drugs,in patients at high cardiovascular risk or previous cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Adults age ≥ 18 years old;
* Patient that could written informed consent;
* Patient with current atherothrombotic cardiovascular disease or at high cardiovascular risk, defined as:
* Patients with previous Coronary Artery Disease (miocardial Infarction, estable or instable angina pectoris or coronary revascularization procedures);
* Patients with previous miocardial Infarction, defined as medical registry (with documentation of at least 2 criterias: clinical symptoms,patological electrocardiogram and elevation of cardiac enzymes- CK-MB and/or troponin);
* Patients with previous brain ischemia (stroke or transient ischemic attack)
* Patients with confirmed previous peripheral arterial disease (Coronary Artery Bypass procedures or angioplasty or amputation due peripheral arterial disease)
* Patients with no established cardiovascular disease but at high cardiovascular risk, defined as 15% or more in 5 years (using the Anderson Framingham scale, 1991)

Exclusion Criteria:

* contraindication for any of the polipill
* If the physician opinion is that terapeutical change could harm the patient (for example, heart failure, need of high beta blocker dose for treatment angina symptons and for the atrial fibrillation rhythm,severe hypertension [degree 3], malignant hypertension or renal insufficiency
* Acute clinical conditions/ surgeries
* Psychiatry clinical conditions(for example, schizophrenia, serious depression)
* pregnant or lactation women
* women at fertile period mulheres not using effective contraceptive methods (oral contraceptive, condom, intrauterine device)
* liver siseases (AST/ALT/FA upon 3 x normal superior limits / bilirrubin upon 1,5 X normal superior limits / diagnosed Liver Cirrhosis
* Renal disfunction (any laboratorial exams upon 3 x normal superior limits)
* Previous participation on other clinical trial
* The participant is unable or refuse to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-10; Primary Completion 2014-04 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
compliance with treatment | 18 months
changed in blood pressure | 18 months
changes in LDL-cholesterol levels | 18 months

SECONDARY OUTCOMES:
the main reason for non compliance with treatment | 18 months
safety of poli pill measures by laboratorial tests | 18 months
  hemogram and blood platelets count, liver function tests (ALT, AST), renal function tests (creatinine).
combined outcome | 18 months
  compound of cardiovascular and total mortality, major cardiovascular events and cholesterol levels.

CONTACTS AND LOCATIONS:
Overall Officials: Otavio Berwanger, PhD, Study Director — Instituto de Ensino e Pesquisa - IEP - HCor
Locations (1):
- Instituto de Ensino e Pesquisa - IEP - HCor, São Paulo, Brazil